CLINICAL TRIAL: NCT02752321
Title: Video Assisted Transitions of Care: The Power of Video for Hospital Discharge Process
Brief Title: An Electronic Multimedia Discharge Application
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: There was a software server issue. Investigators were no longer able to sign patients up to the software program.
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, David Langer, Chairman, Department of Neurosurgery, Lenox Hill Hospital, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 15-260
Record Dates: First submitted 2016-04-15; First posted 2016-04-26 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Hospital Inpatients
Keywords: patient discharge; patient engagement; patient satisfaction; continuity of patient care; hospital discharge; health technology; eDischarge; multimedia; mobile applications; software applications; portable electronic applications
MeSH Terms: conditions — Patient Participation; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- eDischarge + Standard Discharge (SDeD) (Experimental): Patients in this arm will be enrolled in the eDischarge technology prior to hospital discharge. Upon hospital discharge, these patients will receive a personalized eDischarge, containing text and multimedia information, in addition to receiving the standard discharge process.
  Follow-up interviews and surveys will be conducted at 7-14 days post discharge, and at 30-45 days post discharge.
  Interventions: Device: eDischarge
- Standard Discharge (SD) (No Intervention): Patients in this arm will receive the standard discharge process upon hospital discharge.
  Follow-up interviews and surveys will be conducted at 7-14 days post discharge, and at 30-45 days post discharge.

INTERVENTIONS:
Device: eDischarge — Patients will be enrolled in the eDischarge technology during their inpatient hospital stay. A completed electronic discharge packet (EDP) will be given to patients on the day of hospital discharge.
  Arms: eDischarge + Standard Discharge (SDeD)

SUMMARY:
The purpose of this study is to determine whether the addition of a mobile or web based multimedia discharge application (eDischarge) to the discharge process is effective in improving patient experience, engagement, and clinical outcomes in the early post discharge period.

DETAILED DESCRIPTION:
Hospital discharge is an essential transition of a patient's care from the inpatient health care team to the patient and caregiver. While a variety of factors may contribute to the effective discharge process, adequate communication between all parties significantly contributes to better outcomes. However, studies indicate that nearly one in five Medicare patients are re-hospitalized within one month of discharge due to lack of patient understanding and compliance to the post-hospital plan of care.

The standard discharge process, which is similar across all disease etiologies, has not changed significantly in many years and lags behind today's technological advances. Currently, the standard discharge process most commonly is delivered as a written document. This document summarizes the patient's hospitalization and discharge instructions in a plain text format, not significantly personalized, and is reviewed with the patient and caregivers usually at time of the discharge. Patients may not pay attention or understand the clinical information communicated to them and may not remember the dialogues during the discharge. In addition, patients often misplace their discharge papers and will not follow the post discharge instructions.

In early 2009, the Health Information Technology for Economic and Clinical Health (HITECH) Act was adopted to promote the meaningful use of health information technology. Stage 1 of HITECH centered on 5 underlying health outcomes of meaningful use: (1) improve quality, safety, efficiency, and reduce health disparities; (2) engage patients and families in their healthcare; (3) improve care coordination; (4) improve population and public health; and (5) ensure adequate privacy and security protections for personal health information. While the passage of HITECH and application of new database technologies has prompted an increase in the use of electronic health records (EHR), the incentives of meaningful use has not been widely applied (Hsiao and Hing)3.

The current "Age of the Internet" and its ability to deliver data to almost any physical locale instantaneously, including high resolution audio and video, has fostered new ways to create, view and share information - including, potentially, medical records. eDischarge is a new multimedia technology designed to supplement the discharge process and enhance provider-patient communication by facilitating the delivery of discharge and follow-up information to patients. Designed as a secure, HIPPA-compliant, cloud-based software platform, participants are able to access the eDischarge system using a personal computer or a mobile device, which can enhance access to health information for the patient. Through eDischarge, participants are given personalized videos, documents, and images tailored specifically to their particular medical care. eDischarge permits inclusion of both structured health information exchange data as well as medical data to be added to discharge. Providers are able to asynchronously create content throughout a participant's hospital stay, which the participant will be able to access post discharge. The investigators believe that this technology has the potential to improve patient engagement and experience as well as enhance a patient's understanding of his disease process and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ages 18 years and above
* Access to mobile device (phone/tablet) and/or computer at home
* Admission to Lenox Hill Hospital under the Department of Neurosurgery
* Discharge to home and rehab facilities where patients can be accessed

Exclusion Criteria:

* Irreversible impaired brain stem function (bilateral fixed, dilated pupils and extensor motor posturing)
* Patients not expected to survive to the 30 day visit due to co-morbidities or are Do No Resuscitate/Do Not Intubate (DNR/DNI) status prior to randomization
* Patients transferred to a different hospital service or a nursing home
* Patients on hospital precautions or suicide watch, or are deaf or blind
* Any concurrent serious illness that would interfere with the outcome assessments including hepatic, renal, gastroenterologic, respiratory, cardiovascular, endocrinologic, immunologic, and hematologic disease.
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational technology were initiated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2016-08; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Post Discharge Survey | 7-14 Days Post-Discharge
  to determine patient knowledge/awareness of their diagnosis
Post Discharge Survey | 7-14 Days Post-Discharge
  to determine patient knowledge/awareness of their medications

SECONDARY OUTCOMES:
Patient Discharge Experience (eDischarge Questionnaire) | 7-14 Days Post-Discharge
  to compare patients experiences with their discharge between the SDeD and the SD groups.
Patient Discharge Experience (Standard Discharge Questionnaire) | 7-14 Days Post-Discharge
  to compare patients experiences with their discharge between the SDeD and the SD groups.
Hospital Readmission Rate | 30-45 Days Post Discharge
  to compare readmission rates between the SDeD and SD groups.
ED Visit Rate | 30-45 Days Post Discharge
  to compare emergency department visit rates between the SDeD and SD groups.

CONTACTS AND LOCATIONS:
Overall Officials: David J. Langer, MD, Principal Investigator — Northwell Health
Locations (1):
- Lenox Hill Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Forster AJ, Murff HJ, Peterson JF, Gandhi TK, Bates DW. The incidence and severity of adverse events affecting patients after discharge from the hospital. Ann Intern Med. 2003 Feb 4;138(3):161-7. doi: 10.7326/0003-4819-138-3-200302040-00007. PMID 12558354
- [Background] Lai M, Kheterpal S. Creating a real return-on-investment for information system implementation: life after HITECH. Anesthesiol Clin. 2011 Sep;29(3):413-38. doi: 10.1016/j.anclin.2011.05.005. PMID 21871403
- [Background] Hsiao CJ, Hing E. Use and characteristics of electronic health record systems among office-based physician practices: United States, 2001-2013. NCHS Data Brief. 2014 Jan;(143):1-8. PMID 24439138
- [Background] Berkman ND, Dewalt DA, Pignone MP, Sheridan SL, Lohr KN, Lux L, Sutton SF, Swinson T, Bonito AJ. Literacy and health outcomes. Evid Rep Technol Assess (Summ). 2004 Jan;(87):1-8. No abstract available. PMID 15819598